CLINICAL TRIAL: NCT00004797
Title: Pilot Study of Fructose for Sickle Cell Crisis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Shirley Ryan AbilityLab (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11941; NU-573
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Sickle Cell Anemia
Keywords: disease-related problem/condition; genetic diseases and dysmorphic syndromes; hematologic disorders; pain; rare disease; sickle cell anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Genetic Diseases, Inborn; Hematologic Diseases; Pain; Rare Diseases | interventions — Fructose

INTERVENTIONS:
Drug: fructose
Drug: placebo

SUMMARY:
OBJECTIVES: I. Evaluate the efficacy and tolerability of fructose administered every 6 hours for up to 72 hours to patients in active sickle cell crisis.

II. Obtain tolerability information in selected patients treated with fructose for more than 72 hours.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: In the first part of the study, patients are block-randomized (3:1) to a single intravenous dose of fructose or placebo. The dose of fructose is escalated in each successive group after tolerability data are evaluated.

In the second part of the study, patients are randomly assigned (1:1) to fructose or placebo administered intravenously every 6 hours for 72 hours. The dose of fructose is the highest well-tolerated dose determined in Study 1 or the most tolerated dose for the patient. Patients who just completed Study 1 may participate if they are clearly in a separate crisis and continue to meet entry criteria.

Patients whose symptoms persist for more than 72 hours after fructose or placebo are eligible to receive additional fructose every 6 hours until symptoms subside.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Sickle cell crisis requiring hospital admission Crisis began at least 12 hours prior to admission Medical records documenting sickle cell disease and previous crisis requiring hospital visit during the last 24 months available at study site No thalassemia No complex hemoglobinopathy involving thalassemia and sickle cell disease

--Patient Characteristics-- Renal: Creatine no greater than 2.2 mg/dL No requirement for regular dialysis Other: Weight above or below 30% of ideal body weight No fructose intolerance No insulin-dependent diabetes No HIV seropositivity No acquired immune deficiency syndrome (AIDS) or AIDS-related illness No general anesthetic for 7 days prior to and 2 days following entry Primary language allows communication with study staff Demonstration of ability to read and understand pain scales required Ability to identify crisis starting time accurately, i.e., to within 6 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 1995-08

CONTACTS AND LOCATIONS:
Overall Officials: David Green, Study Chair — Shirley Ryan AbilityLab